CLINICAL TRIAL: NCT06553053
Title: Acupuncture Reduces Relapse in Patients With Crohn's Disease: a Superiority Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZYS2024-04
Record Dates: First submitted 2024-08-07; First posted 2024-08-14 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Crohn's Disease Relapse; Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Receiving acupuncture with the function of "harmonizing Shaoyang, nourishing spleen and kidney with warmth"
  Interventions: Other: "Harmonizing Shaoyang, nourishing spleen and kidney with warmth" Acupuncture Group
- Control group (Active Comparator): Receiving acupuncture group with the function of "nourishing spleen and kidney with warmth"
  Interventions: Other: "Nourishing spleen and kidney with warmth" Acupuncture Group

INTERVENTIONS:
Other: "Harmonizing Shaoyang, nourishing spleen and kidney with warmth" Acupuncture Group — Patients receiving acupuncture and mild moxibustion, whom were treated 2 times per week for 12 weeks and followed up for 40 weeks. The first group of acupoints is that CV4 and Bilateral ST37, SP6, SP4, KI3, LI11, SJ4 and GB26 were selected for acupuncture and CV12 and bilateral ST36 and GB41 were selected for moxibustion. The second group of acupoints is that CV12 and Bilateral ST36, GB41, SP4, KI3, LI11, SJ4 and GB26 were selected for acupuncture and CV4 and bilateral SP6 and GB34 were selected for moxibustion. These two groups are alternate. After deqi sensation was even reinforcing and reducing. The surface temperature of acupoints was maintained at 43℃± 1℃ for moxibustion. During each treatment, acupuncture and mild moxibustion are performed simultaneously, both lasting for 30 minutes.
  Arms: Experimental Group
Other: "Nourishing spleen and kidney with warmth" Acupuncture Group — Patients receiving acupuncture and mild moxibustion, whom were treated 2 times per week for 12 weeks and followed up for 40 weeks. The first group of acupoints is that CV4 and Bilateral ST37, SP6, SP4, KI3 and LI11 were selected for acupuncture and CV12 and bilateral ST36 were selected for moxibustion. The second group of acupoints is that CV12 and Bilateral ST36, SP4, KI3 and LI11 were selected for acupuncture and CV4 and bilateral SP6 were selected for moxibustion. These two groups are alternate. After deqi sensation was even reinforcing and reducing. The surface temperature of acupoints was maintained at 43℃± 1℃ for moxibustion. During each treatment, acupuncture and mild moxibustion are performed simultaneously, both lasting for 30 minutes.
  Arms: Control group

SUMMARY:
The aim of this study was to further improve the clinical efficacy of acupuncture in delaying the clinical recurrence of CD and to explore the efficacy mechanism of acupuncture efficacy enhancement.

DETAILED DESCRIPTION:
Acupuncture has been proven to be an effective and safe treatment for CD. In this trial, based on previous studies, which mainly treated CD from the perspective of spleen and stomach tonification, we explored the therapeutic effect of acupuncture in treating CD from the perspective of tonifying the Shaoyang pivot mechanism to enhance the therapeutic effect.Brain-gut axis dysfunction is one of the important pathogenic mechanisms of CD. This trial attempted to explore the therapeutic targets and efficacy mechanisms of acupuncture to enhance CD by analysing brain-gut axis multi-pathway indicators.

ELIGIBILITY:
Inclusion Criteria:

1. patients with clinical diagnosis consistent with CD;
2. aged 16-75;
3. patients in remission (CDAI < 150 and CRP < 5mg/l, or Faecal calprotectin < 50μg/g, or no ulcer under endoscopy);
4. patients with frequent disease recurrences (≥2) in the past years;
5. patients were not taking medication or were only taking one or more of the following drugs: [mesalazine (≤4g/d), prednisone (≤15mg/d), azathioprine (≤1mg/kg/d)] and prednisone and mesalazine were used for at least 1 month, while azathioprine was used for at least 3 months; or those who had poor response or loss of response to biological preparations (anti-TNF-α, IL-12p40, α4β7);
6. those who have never experienced acupuncture;
7. patients signing informed consent.

Exclusion Criteria:

1. patients who are recently pregnant or in pregnancy or lactation;
2. patients with serious organic diseases;
3. patients diagnosed as psychosis;
4. patients who suffer from multiple diseases and need to take other drugs for a long time, and may affect the observation of the efficacy of this trial;
5. severe skin diseases (such as erythema nodosum, pyoderma gangrenosum, etc.), eye diseases (such as iritis, uveitis, etc.), thromboembolic diseases and other serious extraintestinal manifestations;
6. there are serious intestinal fistula, abdominal abscess, intestinal stenosis and obstruction, perianal abscess, gastrointestinal hemorrhage, intestinal perforation and other complications;
7. patients with short bowel syndrome who have undergone abdominal or gastrointestinal surgery in the past half a year;
8. there are skin diseases or defects in the selected area of acupuncture and moxibustion that cannot be performed.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of recurrences | Week 52
  Defined as CDAI > 150 and increase ≥ 70 points, or emergency, hospitalization and surgical events due to worsening of CD conditions, or need to adjust drug to control disease condition.

SECONDARY OUTCOMES:
Number of recurrences | Week 52
  Total number of recurrences. The median number will be counted for both groups.
Time of recurrences | Week 52
  Time to first recurrence will be counted for both groups.
Crohn's disease activity index （CDAI）score | Week 0, 6, 12, 24, 36 and 52
  The mean change in CDAI from baseline. The higher the score, the worse the condition. Greater than 0, no upper limit.
Patient Reported Outcome （PRO2） | Week 0, 6, 12, 24, 36 and 52
  The outcome is measured by level of abdominal pain (visual analogue scale, VAS) and number of diarrhoea in the past week.
First laboratory tests | Week 0, 6, 12, 24, 36 and 52
  serum C-reactive protein (CRP)
Second laboratory tests | Week 0, 6, 12, 24, 36 and 52
  erythrocyte sedimentation rate (ESR)
Third laboratory tests | Week 0, 6, 12, 24, 36 and 52
  platelet count (PLT)
Inflammatory bowel disease questionnaire (IBDQ) | Week 0, 12, 24, 36 and 52
  The mean change in IBDQ from baseline. The higher the score, the worse the condition.The score is range from 32 to 224.
Hospital anxiety and depression scale (HADS) | Week 0, 12, 24, 36 and 52
  The mean change in HADS from baseline. The higher the score, the more serious the disease. The depression and anxiety score is range from 0 to 21.
The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | Week 0, 12, 24, 36 and 52
  The mean change in FACIT-F from baseline. The higher the score, the worse the condition. The score range from 0 to 52.
Colonoscopy or small bowel MR evaluation | Week 0 and 52
  measured by colonoscopy (SES-CD score) or small bowel MR (MaRIA score)
Expectation of acupuncture treatment | Week 0
  measured by acupuncture treatment effectiveness expectation questionnaire
Blind questionnaire | Week 6 and 12
  measured by patients guessing their grouping

OTHER OUTCOMES:
Effects of acupuncture on brain network connectivity properties | Week 0 and 12
  Gray matter structure of the brain，functional connectivity and network properties of brain networks and local activity in brain regions were measured in an attempt to analyze the correlation between changes in these indicators after acupuncture intervention and the efficacy of acupuncture.
Salivary cortisol | Week 0 and 12
  Salivary cortisol is measured by ELISA to analyze effect of acupuncture on HPA axis function.
α-Salivary Amylase | Week 0 and 12
  α-Salivary Amylase is measured by ELISA to analyze effect of acupuncture on HPA axis function.
Serum cortisol | Week 0 and 12
  Serum cortisol is measured by ELISA to analyze effect of acupuncture on HPA axis function.
Effect of acupuncture on autonomic nervous activity | Week 0 and 12
  The effect of acupuncture on autonomic function was recorded by DMS300-4AL.
Effect of acupuncture on intestinal inflammation levels function | Week 0 and 12
  Intestinal inflammation levels are measured by C-reactive protein and plasma concentrations of tumour necrosis factor-α (TNF-α), interleukin-1β (IL-1β), and IL-6.
Effect of acupuncture on intestinal mucosal barrier function | Week 0 and 12
  Intestinal mucosal barrier function are measured by concentrations of lipopolysaccharide (LPS), Diamine oxidase (DAO) and D-lactate.

CONTACTS AND LOCATIONS:
Overall Officials: Bao Chunhui, MD, PhD, Principal Investigator — Shanghai University of TCM
Locations (1):
- Shanghai Research Institute of Acupuncture and Meridian, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dolinger M, Torres J, Vermeire S. Crohn's disease. Lancet. 2024 Mar 23;403(10432):1177-1191. doi: 10.1016/S0140-6736(23)02586-2. Epub 2024 Mar 1. PMID 38437854
- [Background] Roda G, Chien Ng S, Kotze PG, Argollo M, Panaccione R, Spinelli A, Kaser A, Peyrin-Biroulet L, Danese S. Crohn's disease. Nat Rev Dis Primers. 2020 Apr 2;6(1):22. doi: 10.1038/s41572-020-0156-2. PMID 32242028
- [Background] Greuter T, Vavricka SR. Extraintestinal manifestations in inflammatory bowel disease - epidemiology, genetics, and pathogenesis. Expert Rev Gastroenterol Hepatol. 2019 Apr;13(4):307-317. doi: 10.1080/17474124.2019.1574569. Epub 2019 Feb 20. PMID 30791773
- [Background] Ng SC, Leung WK, Shi HY, Li MK, Leung CM, Ng CK, Lo FH, Hui YT, Tsang SW, Chan YK, Loo CK, Chan KH, Hui AJ, Chow WH, Harbord M, Ching JY, Lee M, Chan V, Tang W, Hung IF, Ho J, Lao WC, Wong MT, Sze SF, Shan EH, Lam BC, Tong RW, Mak LY, Wong SH, Wu JC, Chan FK, Sung JJ. Epidemiology of Inflammatory Bowel Disease from 1981 to 2014: Results from a Territory-Wide Population-Based Registry in Hong Kong. Inflamm Bowel Dis. 2016 Aug;22(8):1954-60. doi: 10.1097/MIB.0000000000000846. PMID 27416041
- [Background] Zheng JJ, Zhu XS, Huangfu Z, Gao ZX, Guo ZR, Wang Z. Crohn's disease in mainland China: a systematic analysis of 50 years of research. Chin J Dig Dis. 2005;6(4):175-81. doi: 10.1111/j.1443-9573.2005.00227.x. PMID 16246226
- [Background] Kaplan GG. The global burden of IBD: from 2015 to 2025. Nat Rev Gastroenterol Hepatol. 2015 Dec;12(12):720-7. doi: 10.1038/nrgastro.2015.150. Epub 2015 Sep 1. PMID 26323879
- [Background] Bonovas S, Fiorino G, Allocca M, Lytras T, Nikolopoulos GK, Peyrin-Biroulet L, Danese S. Biologic Therapies and Risk of Infection and Malignancy in Patients With Inflammatory Bowel Disease: A Systematic Review and Network Meta-analysis. Clin Gastroenterol Hepatol. 2016 Oct;14(10):1385-1397.e10. doi: 10.1016/j.cgh.2016.04.039. Epub 2016 May 14. PMID 27189910
- [Background] Esters P, Dignass A. Complementary therapies in inflammatory bowel diseases. Curr Drug Targets. 2014;15(11):1079-88. doi: 10.2174/1389450115666140903112802. PMID 25182607
- [Background] Qu YK, Zhu Y.Differential diagnosis and treatment of Crohn's disease based on the theory of
- [Background] Bao C, Wu L, Wang D, Chen L, Jin X, Shi Y, Li G, Zhang J, Zeng X, Chen J, Liu H, Wu H. Acupuncture improves the symptoms, intestinal microbiota, and inflammation of patients with mild to moderate Crohn's disease: A randomized controlled trial. EClinicalMedicine. 2022 Feb 12;45:101300. doi: 10.1016/j.eclinm.2022.101300. eCollection 2022 Mar. PMID 35198926
- [Background] Gracie DJ, Guthrie EA, Hamlin PJ, Ford AC. Bi-directionality of Brain-Gut Interactions in Patients With Inflammatory Bowel Disease. Gastroenterology. 2018 May;154(6):1635-1646.e3. doi: 10.1053/j.gastro.2018.01.027. Epub 2018 Jan 31. PMID 29366841
- [Background] Gracie DJ, Hamlin PJ, Ford AC. The influence of the brain-gut axis in inflammatory bowel disease and possible implications for treatment. Lancet Gastroenterol Hepatol. 2019 Aug;4(8):632-642. doi: 10.1016/S2468-1253(19)30089-5. Epub 2019 May 20. PMID 31122802
- [Background] Fairbrass KM, Lovatt J, Barberio B, Yuan Y, Gracie DJ, Ford AC. Bidirectional brain-gut axis effects influence mood and prognosis in IBD: a systematic review and meta-analysis. Gut. 2022 Sep;71(9):1773-1780. doi: 10.1136/gutjnl-2021-325985. Epub 2021 Nov 1. PMID 34725197
- [Background] Pellissier S, Dantzer C, Mondillon L, Trocme C, Gauchez AS, Ducros V, Mathieu N, Toussaint B, Fournier A, Canini F, Bonaz B. Relationship between vagal tone, cortisol, TNF-alpha, epinephrine and negative affects in Crohn's disease and irritable bowel syndrome. PLoS One. 2014 Sep 10;9(9):e105328. doi: 10.1371/journal.pone.0105328. eCollection 2014. PMID 25207649
- [Background] Bonaz B, Sinniger V, Hoffmann D, Clarencon D, Mathieu N, Dantzer C, Vercueil L, Picq C, Trocme C, Faure P, Cracowski JL, Pellissier S. Chronic vagus nerve stimulation in Crohn's disease: a 6-month follow-up pilot study. Neurogastroenterol Motil. 2016 Jun;28(6):948-53. doi: 10.1111/nmo.12792. Epub 2016 Feb 27. PMID 26920654
- [Background] Tillisch K, Labus JS. Advances in imaging the brain-gut axis: functional gastrointestinal disorders. Gastroenterology. 2011 Feb;140(2):407-411.e1. doi: 10.1053/j.gastro.2010.12.014. Epub 2010 Dec 15. No abstract available. PMID 21167161
- [Background] Stasi C, Orlandelli E. Role of the brain-gut axis in the pathophysiology of Crohn's disease. Dig Dis. 2008;26(2):156-66. doi: 10.1159/000116774. Epub 2008 Apr 21. PMID 18431066
- [Background] del Rey A, Klusman I, Besedovsky HO. Cytokines mediate protective stimulation of glucocorticoid output during autoimmunity: involvement of IL-1. Am J Physiol. 1998 Oct;275(4):R1146-51. doi: 10.1152/ajpregu.1998.275.4.R1146. PMID 9756545
- [Background] Mackner LM, Clough-Paabo E, Pajer K, Lourie A, Crandall WV. Psychoneuroimmunologic factors in inflammatory bowel disease. Inflamm Bowel Dis. 2011 Mar;17(3):849-57. doi: 10.1002/ibd.21430. Epub 2010 Aug 18. PMID 20722061
- [Background] Wang L, Bai AP. Dysfunction of the autonomic nervous system and inflammatory bowel disease.World Chinese Journal of Digestology 2012;[20]20: 3010-3014.
- [Background] Pellissier S, Dantzer C, Canini F, Mathieu N, Bonaz B. Psychological adjustment and autonomic disturbances in inflammatory bowel diseases and irritable bowel syndrome. Psychoneuroendocrinology. 2010 Jun;35(5):653-62. doi: 10.1016/j.psyneuen.2009.10.004. Epub 2009 Nov 11. PMID 19910123
- [Background] Prame Kumar K, Ooi JD, Goldberg R. The interplay between the microbiota, diet and T regulatory cells in the preservation of the gut barrier in inflammatory bowel disease. Front Microbiol. 2023 Dec 1;14:1291724. doi: 10.3389/fmicb.2023.1291724. eCollection 2023. PMID 38107848
- [Background] Bao CH, Liu P, Liu HR, Wu LY, Shi Y, Chen WF, Qin W, Lu Y, Zhang JY, Jin XM, Wang XM, Zhao JM, Liu XM, Tian J, Wu HG. Alterations in brain grey matter structures in patients with crohn's disease and their correlation with psychological distress. J Crohns Colitis. 2015 Jul;9(7):532-40. doi: 10.1093/ecco-jcc/jjv057. Epub 2015 Apr 20. PMID 25895879
- [Background] Bao CH, Liu P, Liu HR, Wu LY, Jin XM, Wang SY, Shi Y, Zhang JY, Zeng XQ, Ma LL, Qin W, Zhao JM, Calhoun VD, Tian J, Wu HG. Differences in regional homogeneity between patients with Crohn's disease with and without abdominal pain revealed by resting-state functional magnetic resonance imaging. Pain. 2016 May;157(5):1037-1044. doi: 10.1097/j.pain.0000000000000479. PMID 26761381
- [Background] Agostini A, Benuzzi F, Filippini N, Bertani A, Scarcelli A, Farinelli V, Marchetta C, Calabrese C, Rizzello F, Gionchetti P, Ercolani M, Campieri M, Nichelli P. New insights into the brain involvement in patients with Crohn's disease: a voxel-based morphometry study. Neurogastroenterol Motil. 2013 Feb;25(2):147-e82. doi: 10.1111/nmo.12017. Epub 2012 Sep 23. PMID 22998431
- [Background] Bao CH, Xu S, Wu LY, et al. Brain imaging features predict disease activity in patients with Crohn's disease. Gastroenterology, 2024, 166(5): S-205.
- [Background] Bao CH, Wu LY, Liu HR, et al. Acupuncture reduces clinical relapse in Crohn's disease: a randomized controlled trial. Gastroenterology, 2023, 164(6): S-1093.
- [Background] Chow, S.C., Shao, J., and Wang, H. 2008. Sample Size Calculations in Clinical Research, Second Edition.Chapman & Hall/CRC. Boca Raton, Florida.
- [Background] Inflammatory Bowel Disease Group, Chinese Society of Gastroenterology Chinese Medical Association, Inflammatory Bowel Disease Quality Control Center of China.Chinese clinical practice guideline on the management of Crohn's disease (2023, Guangzhou)[J].Chinese Journal of Inflammatory Bowel Diseases, 2024,8(1):2-32.
- [Background] Albenberg L, Brensinger CM, Wu Q, Gilroy E, Kappelman MD, Sandler RS, Lewis JD. A Diet Low in Red and Processed Meat Does Not Reduce Rate of Crohn's Disease Flares. Gastroenterology. 2019 Jul;157(1):128-136.e5. doi: 10.1053/j.gastro.2019.03.015. Epub 2019 Mar 11. PMID 30872105